CLINICAL TRIAL: NCT06120621
Title: Combined Visco-Circumferential-Suture-Trabeculotomy With Phacoemulsification Versus Phacoemulsification in Primary Angle Closure Glaucoma: A 2-Year Randomized Controlled Trial.
Brief Title: Combined VCST With Phacoemulsification Versus Phacoemulsification in Primary Angle Closure Glaucoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Dina abdelfattah, lecturer of ophthalmology , Faculty of medicine, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R.23.10.2345.R1
Record Dates: First submitted 2023-10-24; First posted 2023-11-07 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Narrow-Angle Glaucoma
MeSH Terms: conditions — Glaucoma, Angle-Closure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Active Comparator): Visco-Circumferential-Suture-Trabeculotomy followed by Phacoemulsification
  Interventions: Procedure: Arm 1 : VCST-phaco group , Arm 2 : phaco group.
- Arm 2 (Active Comparator): phacoemulsification alone
  Interventions: Procedure: Arm 1 : VCST-phaco group , Arm 2 : phaco group.

INTERVENTIONS:
Procedure: Arm 1 : VCST-phaco group , Arm 2 : phaco group. — Arm 1 : VCST-phaco group , Arm 2 : phaco group.

SUMMARY:
As ab externo metal probe trabeculotomy cannot achieve 360-degree circumferential angle surgery, prolene suture can be used to achieve this without the need for an illuminated microcatheter. In order to combine the advantages of the use of viscoelastic and those of circumferential trabeculotomy, this technique (Visco-Circumferential-Suture- Trabeculotomy "VCST") was previously used successfully in PCG. In the current study , the authors hypothesize that combination of VCST with phacoemulsification in primary angle closure glaucoma patients may have an added affect to phacoemulsification alone in cases with more extent of angle damage and that the injection of a viscoelastic into both ends of the unroofed SC before its cannulation by a polypropylene suture and subsequent circumferential trabeculotomy may facilitate circumferential cannulation of SC and hence the trabeculotomy and increase the success of the technique

DETAILED DESCRIPTION:
Aim of the work: To assess the surgical outcomes of Combined Visco-Circumferential-Suture-Trabeculotomy with Phacoemulsification compared to phacoemulsification alone in the management of chronic primary angle closure glaucoma (CPACG).

Patients & Methods:

This is a prospective randomized controlled clinical trial including eyes with uncontrolled CPACG and indicated for surgery. The study will be held in Mansoura ophthalmic center in the duration from September 2023 and March 2024. Patients will be randomized to undergo either Visco-Circumferential-Suture-Trabeculotomy followed by Phacoemulsification (VCST-phaco group) or phacoemulsification alone (phaco group). Randomization will be done through closed envelope method.

Sample size was calculated using website, http://www.raosoft.com/samplesize.html Values for prevalence of primary angle closure glaucoma were used to calculate the study population from Cheng et al. 50 cases will be included in the study, 25 for each group Patients will be included in the study if they have (1) PACG (2) a patent iridotomy, (3) synechial angle closure of more than 180 degrees that occluded the trabecular meshwork as confirmed by indentation gonioscopy, (4) an IOP greater than 21 mm Hg despite maximally tolerated antiglaucoma medications, and (5) no history of intraocular surgery other than laser iridotomy. Primary ACG is defined by the presence of elevated IOP (>21 mm Hg) and synechial angle closure of a gonioscopically narrow angle with optic nerve cupping typical of glaucoma and corresponding matching visual field defects. Patients with an acute attack or a known recent chronic ACG attack will be excluded from the study. Patients with primary open-angle glaucoma and secondary glaucomas who are on anticoagulant therapy and cannot stop treatment or with media opacity that interfere with cataract surgery, visual field testing, or OCT imaging will be excluded from the study.

In all patients, a thorough history will be taken then a full ophthalmological examination will be done, particularly estimation of the best corrected visual acuity (BCVA) using the decimal notation, slit lamp examination, and IOP measurement by Goldmann's applanation tonometry. Gonioscopy using Goldmann 3-mirrors goniolens for angle grading using Schaffer's grading system and fundus examination. Visual field (VF) assessment will be performed by SITA strategy perimetry (Humphrey, central 24-2 standard strategy). Retinal nerve fiber layer (RNFL) thickness and optic nerve head will be evaluated using a spectral domain optical coherence tomography (OCT; Topcon, Japan). Ultrasound biometry will be performed, and the anterior chamber depth (ACD) will be recorded. The number of antiglaucoma medications is also recorded.

Postoperative follow up visits will be planned on the first day, first week, second week, at first month, three months and six months. Outcome measures include the IOP value at each visit, BCVA, the number of IOP lowering medications used, and occurrence of any complications. The criteria for complete success is defined as an intraocular pressure between 6 and 18 mmHg, with a reduction of at least 30% from the baseline IOP. This should be achieved without the use of IOP-lowering medications or further surgery and any vision-threatening complications. Qualified success is defined as the same criteria for complete success but with the use of IOP-lowering medications.

ELIGIBILITY:
Inclusion Criteria:patients with:

* PACG
* patent iridotomy,
* synechial angle closure of more than 180 degrees that occluded the trabecular meshwork as confirmed by indentation gonioscopy
* an IOP greater than 21 mm Hg despite maximally tolerated antiglaucoma medications -no history of intraocular surgery other than laser iridotomy. -

Exclusion Criteria:

* Patients with primary open-angle glaucoma
* secondary glaucomas
* patients on anticoagulant therapy and cannot stop treatment
* patients with media opacity that interfere with cataract surgery, visual field testing, or OCT imaging

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
IOP control | one year
  The criteria for complete success is defined as an intraocular pressure between 6 and 18 mmHg, with a reduction of at least 30% from the baseline IOP. This should be achieved without the use of IOP-lowering medications or further surgery and any vision-threatening complications. Qualified success is defined as the same criteria for complete success but with the use of IOP-lowering medications.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed El wehidy, professor, Principal Investigator — professor of ophthalmology, Mansoura university
Locations (1):
- Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
results will be shared